CLINICAL TRIAL: NCT05576714
Title: Investigation of Prognostic Biomarkers, Host Factors and Viral Factors for COVID-19 Associated Encephalopathy/Encephalitis and Multi-systemic Inflammatory Syndrome in Children
Brief Title: Investigation of Prognostic Biomarkers, Host Factors and Viral Factors for COVID-19 in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Medical Foundation (Other); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Mackay Memorial Hospital (Other); Tri-Service General Hospital (Other); National Health Research Institutes, Taiwan (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 202207201RIND
Record Dates: First submitted 2022-10-10; First posted 2022-10-12 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: COVID-19-Associated Encephalitis; Multisystem Inflammatory Syndrome in Children
Keywords: COVID-19; encephalitis; MIS-C
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19; Encephalitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood, nasopharyngeal swab, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- encephalopathy/encephalitis: Children will be classified as the following four diagnoses: 1. Encephalopathy (MERS, ANEC, ASED); 2. Acute encephalitis; 3. ADEM; 4. Fulminant cerebral edema. The classification will be adjudicated and discussed by neurology and critical care experts on the NTUH and CGMH study team (W.T.L, J.J.L, and K.L.L.)
  Interventions: Other: delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis
- MIS-C: The following 6 criteria for MIS-C have to be met: age 0 to 19 years, fever for ≥3 days, clinical signs of multisystem involvement (at least 2 systems), elevated markers of inflammation (e.g., CRP, procalcitonin or ferritin), evidence of SARS-CoV-2 infection and no other obvious microbial cause of inflammation.
  Interventions: Other: delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis
- control group: Age and gender matched healthy control children or mild COVID-19 cases without MIS-C will be also included for further comparison
  Interventions: Other: delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis

INTERVENTIONS:
Other: delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis — We will delineate the clinical and laboratory characteristics of COVID-19 associated encephalopathy and encephalitis, the role of immune, virology, genetics mechanism in pathophysiology, and will optimize the treatment algorithm based on the result of this study. We also expect that the important biomarkers and risk factors associated with clinical outcome and severity, the immunopathogenesis of MIS-C, host genetic factors and the viral pathogenesis and microbiota associated with MIS-C will be found.

SUMMARY:
Background and objective From this April, there was a COVID-19 outbreak in Taiwan. The first fatal case of pediatric COVID-19 encephalitis was reported on April 19, 2022 and fatal fulminant cerebral edema in other 4 children with COVID-19 encephalitis was reported within 1 month from Taiwan CDC registry. To date, around 700,000 children got COVID-19 recently. Several children developed MIS-C (multi-system inflammatory syndrome in children)-related shock about 2-6 weeks after COVID-19. Since both COVID-19 associated encephalopathy/ encephalitis and MIS-C are life-threatening, it is urgent to delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis.

Methods Pediatricians will enroll cases of both COVID-19 associated encephalopathy/ encephalitis and MIS-C from several hospitals and medical centers. Their clinical manifestations, lab findings, severity and outcomes will be collected. Clinical assessment of all the systems will be performed. Blood, nasopharyngeal swab and stool will be collected at acute, subacute and convalescent stages for whole exome sequencing, immunopathogenesis including chemokine/cytokine, T/B lymphocyte subset, SARS-CoV2 specific Ab/T/B cell, T and B cell repertoire, viral pathogenesis including multiple viral detection, persistence of fecal SARS-COVID-2 as well as respiratory and gut microbiota. We will establish the animal models for COVID-19 associated encephalopathy/encephalitis and MIS-C, based on the K18-hACE2 or R26R-AGP mouse models established in NTU animal center. Moreover, specific viral or host factors involved in regulating the pathogenesis and immune responses can be investigated, to optimize the protocol for further improvement of the animal models and also to help identify the putative therapeutic targets.

Expected results We will delineate the clinical and laboratory characteristics of COVID-19 associated encephalopathy and encephalitis, the role of immune, virology, genetics mechanism in pathophysiology, and will optimize the treatment algorithm based on the result of this study. We also expect that the important biomarkers and risk factors associated with clinical outcome and severity, the immunopathogenesis of MIS-C, host genetic factors and the viral pathogenesis and microbiota associated with MIS-C will be found.

DETAILED DESCRIPTION:
Background for COVID-19 associated encephalopathy/encephalitis in children The COVID-19 primarily cause the respiratory diseases, such as croup, bronchiolitis, or pneumonia, but it also can affect the nervous system. According to the data of 1,695 children and adolescents, from March 15, 2020, to December 15, 2020, hospitalized for COVID-19 in 61 hospitals in the United States, 365 (22%) were found to have neurological symptoms. The majority children (322 children, 88%) had transient neurological symptoms. Unfortunately, 43 of them (12%) developed severe life-threatening conditions, including severe encephalopathy (15 children), ischemia or hemorrhagic stroke (12 children), acute central nervous system infection or acute disseminated encephalomyelitis (ADEM) (8 children), acute fulminant cerebral edema (4 children), and Guillain-Barré syndrome (GBS) (4 children). Of the 43 children, 11 patients (26%) died, and another 40% were discharged from the hospital with new neurological sequelae. In Asia, Hong Kong also experienced the Omicron pandemic in March. 171 (14.9%) of 1147 children hospitalized for Omicron were found to have neurological manifestations. The most common was the febrile seizure (11.60%), but there were also 5 children (0.44%) who developed coronavirus-related encephalopathy or encephalitis. Finally, two of them died of neurological causes: one with encephalopathy and the other with fulminant cerebral oedema.

Although the clinical course of acute encephalitis caused by COVID-19 in children is relatively mild in United States and European, the clinical course seemed to be more severe and fulminant in Taiwan. There are five cases of COVID-19 associated encephalopathy and encephalitis in Hong Kong, but the data available for reference is limited. Besides, the clinical course and pathophysiology of children with COVID-19 associated encephalopathy and encephalitis in Taiwan were unknown, it urgently need a clinically oriented, integrated research project.

Clinical research projects for COVID-19 associated encephalopathy/encephalitis in children The aim of this project is

1. To analyze the clinical course and classify the stage of COVID-19 associated encephalopathy and encephalitis in children 2. To find the clinical predictor, biomarker, and imaging characteristic in critical case of COVID-19 associated encephalopathy and encephalitis in children 3. To explore the immune mechanism of COVID-19 associated encephalopathy and encephalitis in children 4. To explore the role of genetics in COVID-19 associated encephalopathy and encephalitis in children 5.To Explore the role of viral variants and co-infection in COVID-19 associated encephalopathy and encephalitis in children 6. To establish proper animal models for studying the pathogenesis and therapeutics for COVID-19 associated encephalopathy/encephalitis

Method: case planning for COVID-19 associated encephalopathy/encephalitis in children Active surveillance will be performed nationally to identify children and adolescents (age≤18 years) with COVID-19 related illness hospitalized from July 01, 2022, to February 28, 2023. The data will registry to the public database hold by NTUH and CGMH.

Estimated including patient number:

110 children (critical group: 30 children; non-critical group:80 children) Including criteria

1. Age less than 18 years old.
2. A positive SARS-CoV-2 test result (reverse transcriptase-polymerase chain reaction and/or antibody)。
3. Hospitalized children.
4. Clinical diagnostic criteria for encephalitis.

   Major criteria:
   1. . Altered mental status greater than 24 hours without alternative cause identified Minor criteria: need at least 2 minor criteria for encephalitis

   <!-- -->

   1. Fever
   2. Seizures
   3. Focal neurologic signs
   4. CSF: pleocytosis
   5. EEG: abnormal slow background or epileptiform discharge
   6. Neuroimaging: abnormal brain inflammation on MRI *****Major+2 minor: possible encephalitis; Major+3 minor: probable encephalitis; Brain biopsy: confirmed encephalitis Exclusion criteria

   1) Age more than 18 years old 2) Previous history of encephalopathy, acute encephalopathy caused by other etiology, not COVID-19, development delay, autism, ADHD, epilepsy and febrile seizure 3) Non-hospitalized children Critical case was defined as children who admitted to pediatric intensive care unit. And Non-critical case was defined as children who admitted to general ward.

   Classification of COVID-19 associated encephalopathy and encephalitis Children will be classified as the following four diagnoses: 1. Encephalopathy (MERS, ANEC, ASED); 2. Acute encephalitis; 3. ADEM; 4. Fulminant cerebral edema. The classification will be adjudicated and discussed by neurology and critical care experts on the NTUH and CGMH study team (W.T.L, J.J.L, and K.L.L.)

   Method: Research content for COVID-19 associated encephalopathy/encephalitis in children Clinical manifestations and laboratory/imaging data collection This is a prospective observational study that does not involve clinical treatment. We propose a schedule for specimen collection /examination in clinical care. The routine ICU laboratory test on day 1, 2,3 7 include CBC/DC, PT/APTT, Fibrinogen, d-dimer, AST/ALT, BUN/Cr, Troponin-I, CPK, BNP or NT-Pro-BNP, CK-MB, Na/K/Cl/Ca/P/Mg, cholesterol, TG, CRP, PCT, IL-6, Ferritin, LDH. We also collect the serum before immunotherapy (such as IVIG, IL-6 antagonist (Tocilizumab) or methylprednisolone pulse therapy) and PMBC (peripheral blood mononuclear cell). Besides, throat swab, Filmarray NP panel (depends on the situation of each hospital) will be also arranged. If lumbar puncture will be performed, routine CSF survey will include routine (WBC)/biochemistry (TP, sugar, lactate)/culture/Filmarray ME panel and 1 ml of CSF will be also reverse. In term of examination, EEG, brain CT and/or MRI will also encourage and depend on the situation of each hospital. Besides, we will also perform the 2D echo and EKG for evaluation of cardiac function of these patients.

   We will perform systematic data collection, including past history (such as preterm, congenital heart disease, chronic lung disease, obesity and DM), the evolution of the disease course, the results of routine clinical tests and examinations and outcome. The disease course includes the worse vital signs of every day, time to start use of antivirus drug, immunotherapy, inotropic agent, ventilator, anticonvulsant and IICP management. Outcomes will be determined at hospital discharge. The primary outcome is mortality. The secondary outcome is ICU stay, duration of hospitalization and neurologic outcome. Neurologic deficits are defined as gross impairment in motor, cognitive, or speech and language functions as well as epilepsy.

   Background for MIS-C From this April, there was a big COVID-19 outbreak in Taiwan. Infection with COVID-19 was laboratory-confirmed in 3,803,049 cases and about 20% of the cases were children, so around 700,000 children got COVID-19 recently in Taiwan. Several children developed MIS-C (multi-system inflammatory syndrome in children)-related shock about 1 month after COVID-19. There would be about 200 MIS-C in Taiwan if the incidence of MIS-C per 1,000,000 COVID-19 infections is around 300 according to the recent reports. Since MIS-C is life-threatening, it is urgent to delineate its prognostic biomarker, host genetic factors, immunopathogenesis and viral pathogenesis.

   The study flow chart of MIS-C is the following:

   (1). TPIDA Clinical core for Case enrollment, data and sample collection The clinical study will be conducted by Taiwan Pediatric Infectious Disease Alliance (TPIDA), a collaborative consortium of pediatric infectious disease departments in tertiary medical centers in Taiwan.

   A. Pediatricians of TPIDA will enroll 100 to 200 cases of MIS-C at National Taiwan University Children Hospital, Chang Gung Memorial Hospital, National Taiwan University Hospital Hsin-Chu Branch and Yun-Lin Branch, Chi-Mei Medical Center, National Cheng Gung University Hospital and MacKay Children Hospital after the written informed consent is obtained from their parents or guardians. The following 6 criteria for MIS-C have to be met: age 0 to 19 years, fever for ≥3 days, clinical signs of multisystem involvement (at least 2 systems), elevated markers of inflammation (e.g., CRP, procalcitonin or ferritin), evidence of SARS-CoV-2 infection and no other obvious microbial cause of inflammation.

   B. Clinical severity The severity of MIS-C will be dependent on the degree of inflammation, heart involvement and the presence of shock. Mild MIS-C is defined as without shock, moderate as shock with VIS score less than 10, and severe as shock with VIS score equal or over 10. [Vasoactive-Inotropic Score (VIS) = Dopamine dose (μg/kg/min) + Dobutamine dose (μg/kg/min) + 10 x Milrinone dose (μg/kg/min) + 100 x Epinephrine dose (μg/kg/min) + 100 x Norepinephrine dose (μg/kg/min) + 10,000 x Vasopressin dose (units/kg/min)].

   C. Clinical assessment and data collection Demographics, BMI, underlying medical diseases, past history of hospitalization and COVID-19 infection, past history or family history of Kawasaki disease, COVID-19 vaccination status, and their current clinical manifestations such as fever, mucocutaneous manifestations, lymphadenopathy, gastrointestinal symptoms, activity, appetite, urine output, treatment including intravenous immunoglobulin (IVIG), steroid, immunomodulators, inotropic agents, antibiotics and outcome will be collected.

   D. Sample collection For the subsequent workup of viral pathogenesis, host genetic factors and immunopathogenesis, the following specimens will be collected at different stages.

   E. Control group Age and gender matched healthy control children or mild COVID-19 cases without MIS-C will be also included for further comparison.

   F. Retrospective and prospective case review The clinical manifestations, lab findings, severity, treatment and outcomes of the MIS-C cases, either retrospectively collected or prospectively enrolled, will be collected and analyzed to find the important biomarkers and risk factors associated with their clinical severity and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 18 years old.
2. A positive SARS-CoV-2 test result (reverse transcriptase-polymerase chain reaction and/or antibody)。
3. Hospitalized children.
4. Clinical diagnostic criteria for encephalitis.

Major criteria:

1). Altered mental status greater than 24 hours without alternative cause identified Minor criteria: need at least 2 minor criteria for encephalitis

1. Fever
2. Seizures
3. Focal neurologic signs
4. CSF: pleocytosis
5. EEG: abnormal slow background or epileptiform discharge
6. Neuroimaging: abnormal brain inflammation on MRI *****Major+2 minor: possible encephalitis; Major+3 minor: probable encephalitis; Brain biopsy: confirmed encephalitis

The following 6 criteria for MIS-C have to be met: age 0 to 19 years, fever for ≥3 days, clinical signs of multisystem involvement (at least 2 systems), elevated markers of inflammation (e.g., CRP, procalcitonin or ferritin), evidence of SARS-CoV-2 infection and no other obvious microbial cause of inflammation.

Exclusion Criteria:

1. Age more than 18 years old
2. Previous history of encephalopathy, acute encephalopathy caused by other etiology, not COVID-19, development delay, autism, ADHD, epilepsy and febrile seizure
3. Non-hospitalized children

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Active surveillance will be performed nationally to identify children and adolescents (age≤18 years) with COVID-19 related illness hospitalized from July 01, 2022, to February 28, 2023. The data will registry to the public database hold by NTUH and CGMH.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
clinical and laboratory characteristics of COVID-19 associated encephalitis/encephalopathy | 2 year
  for example: fever, poor consciousness, persistent lethargy, persistent headache, persistent vomiting, muscle twitching, convulsions, unsteady gait, etc.
biomarkers and risk factors of MIS-C | 2 year
  the immunopathogenesis of MIS-C, host genetic factors and the viral pathogenesis and microbiota associated with MIS-C will be found.

CONTACTS AND LOCATIONS:
Overall Officials: Luna-Yin Chang, professor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Chung Cheng District, Taiwan

REFERENCES:
- [Background] Nygaard U, Holm M, Hartling UB, Glenthoj J, Schmidt LS, Nordly SB, Matthesen AT, von Linstow ML, Espenhain L. Incidence and clinical phenotype of multisystem inflammatory syndrome in children after infection with the SARS-CoV-2 delta variant by vaccination status: a Danish nationwide prospective cohort study. Lancet Child Adolesc Health. 2022 Jul;6(7):459-465. doi: 10.1016/S2352-4642(22)00100-6. Epub 2022 May 6. PMID 35526537
- [Background] Payne AB, Gilani Z, Godfred-Cato S, Belay ED, Feldstein LR, Patel MM, Randolph AG, Newhams M, Thomas D, Magleby R, Hsu K, Burns M, Dufort E, Maxted A, Pietrowski M, Longenberger A, Bidol S, Henderson J, Sosa L, Edmundson A, Tobin-D'Angelo M, Edison L, Heidemann S, Singh AR, Giuliano JS Jr, Kleinman LC, Tarquinio KM, Walsh RF, Fitzgerald JC, Clouser KN, Gertz SJ, Carroll RW, Carroll CL, Hoots BE, Reed C, Dahlgren FS, Oster ME, Pierce TJ, Curns AT, Langley GE, Campbell AP; MIS-C Incidence Authorship Group; Balachandran N, Murray TS, Burkholder C, Brancard T, Lifshitz J, Leach D, Charpie I, Tice C, Coffin SE, Perella D, Jones K, Marohn KL, Yager PH, Fernandes ND, Flori HR, Koncicki ML, Walker KS, Di Pentima MC, Li S, Horwitz SM, Gaur S, Coffey DC, Harwayne-Gidansky I, Hymes SR, Thomas NJ, Ackerman KG, Cholette JM. Incidence of Multisystem Inflammatory Syndrome in Children Among US Persons Infected With SARS-CoV-2. JAMA Netw Open. 2021 Jun 1;4(6):e2116420. doi: 10.1001/jamanetworkopen.2021.16420. PMID 34110391
- [Background] Ghosh P, Katkar GD, Shimizu C, Kim J, Khandelwal S, Tremoulet AH, Kanegaye JT; Pediatric Emergency Medicine Kawasaki Disease Research Group; Bocchini J, Das S, Burns JC, Sahoo D. An Artificial Intelligence-guided signature reveals the shared host immune response in MIS-C and Kawasaki disease. Nat Commun. 2022 May 16;13(1):2687. doi: 10.1038/s41467-022-30357-w. PMID 35577777
- [Background] Chou J, Platt CD, Habiballah S, Nguyen AA, Elkins M, Weeks S, Peters Z, Day-Lewis M, Novak T, Armant M, Williams L, Rockowitz S, Sliz P, Williams DA, Randolph AG, Geha RS; Taking on COVID-19 Together Study Investigators. Mechanisms underlying genetic susceptibility to multisystem inflammatory syndrome in children (MIS-C). J Allergy Clin Immunol. 2021 Sep;148(3):732-738.e1. doi: 10.1016/j.jaci.2021.06.024. Epub 2021 Jul 2. PMID 34224783
- [Background] Sacco K, Castagnoli R, Vakkilainen S, Liu C, Delmonte OM, Oguz C, Kaplan IM, Alehashemi S, Burbelo PD, Bhuyan F, de Jesus AA, Dobbs K, Rosen LB, Cheng A, Shaw E, Vakkilainen MS, Pala F, Lack J, Zhang Y, Fink DL, Oikonomou V, Snow AL, Dalgard CL, Chen J, Sellers BA, Montealegre Sanchez GA, Barron K, Rey-Jurado E, Vial C, Poli MC, Licari A, Montagna D, Marseglia GL, Licciardi F, Ramenghi U, Discepolo V, Lo Vecchio A, Guarino A, Eisenstein EM, Imberti L, Sottini A, Biondi A, Mato S, Gerstbacher D, Truong M, Stack MA, Magliocco M, Bosticardo M, Kawai T, Danielson JJ, Hulett T, Askenazi M, Hu S; NIAID Immune Response to COVID Group; Chile MIS-C Group; Pavia Pediatric COVID-19 Group; Cohen JI, Su HC, Kuhns DB, Lionakis MS, Snyder TM, Holland SM, Goldbach-Mansky R, Tsang JS, Notarangelo LD. Immunopathological signatures in multisystem inflammatory syndrome in children and pediatric COVID-19. Nat Med. 2022 May;28(5):1050-1062. doi: 10.1038/s41591-022-01724-3. Epub 2022 Feb 17. PMID 35177862
- [Background] Kumar D, Rostad CA, Jaggi P, Villacis Nunez DS, Prince C, Lu A, Hussaini L, Nguyen TH, Malik S, Ponder LA, Shenoy SPV, Anderson EJ, Briones M, Sanz I, Prahalad S, Chandrakasan S. Distinguishing immune activation and inflammatory signatures of multisystem inflammatory syndrome in children (MIS-C) versus hemophagocytic lymphohistiocytosis (HLH). J Allergy Clin Immunol. 2022 May;149(5):1592-1606.e16. doi: 10.1016/j.jaci.2022.02.028. Epub 2022 Mar 15. PMID 35304157
- [Background] Sharma C, Ganigara M, Galeotti C, Burns J, Berganza FM, Hayes DA, Singh-Grewal D, Bharath S, Sajjan S, Bayry J. Multisystem inflammatory syndrome in children and Kawasaki disease: a critical comparison. Nat Rev Rheumatol. 2021 Dec;17(12):731-748. doi: 10.1038/s41584-021-00709-9. Epub 2021 Oct 29. PMID 34716418
- [Background] Natarajan A, Zlitni S, Brooks EF, Vance SE, Dahlen A, Hedlin H, Park RM, Han A, Schmidtke DT, Verma R, Jacobson KB, Parsonnet J, Bonilla HF, Singh U, Pinsky BA, Andrews JR, Jagannathan P, Bhatt AS. Gastrointestinal symptoms and fecal shedding of SARS-CoV-2 RNA suggest prolonged gastrointestinal infection. Med. 2022 Jun 10;3(6):371-387.e9. doi: 10.1016/j.medj.2022.04.001. Epub 2022 Apr 13. PMID 35434682
- [Background] Yonker LM, Gilboa T, Ogata AF, Senussi Y, Lazarovits R, Boribong BP, Bartsch YC, Loiselle M, Rivas MN, Porritt RA, Lima R, Davis JP, Farkas EJ, Burns MD, Young N, Mahajan VS, Hajizadeh S, Lopez XIH, Kreuzer J, Morris R, Martinez EE, Han I, Griswold K Jr, Barry NC, Thompson DB, Church G, Edlow AG, Haas W, Pillai S, Arditi M, Alter G, Walt DR, Fasano A. Multisystem inflammatory syndrome in children is driven by zonulin-dependent loss of gut mucosal barrier. J Clin Invest. 2021 Jul 15;131(14):e149633. doi: 10.1172/JCI149633. PMID 34032635
- [Background] Diorio C, Shraim R, Vella LA, Giles JR, Baxter AE, Oldridge DA, Canna SW, Henrickson SE, McNerney KO, Balamuth F, Burudpakdee C, Lee J, Leng T, Farrel A, Lambert MP, Sullivan KE, Wherry EJ, Teachey DT, Bassiri H, Behrens EM. Proteomic profiling of MIS-C patients indicates heterogeneity relating to interferon gamma dysregulation and vascular endothelial dysfunction. Nat Commun. 2021 Dec 10;12(1):7222. doi: 10.1038/s41467-021-27544-6. PMID 34893640
- [Background] Qian Y, Lei T, Patel PS, Lee CH, Monaghan-Nichols P, Xin HB, Qiu J, Fu M. Direct Activation of Endothelial Cells by SARS-CoV-2 Nucleocapsid Protein Is Blocked by Simvastatin. J Virol. 2021 Nov 9;95(23):e0139621. doi: 10.1128/JVI.01396-21. Epub 2021 Sep 22. PMID 34549987
- [Background] Oladunni FS, Park JG, Pino PA, Gonzalez O, Akhter A, Allue-Guardia A, Olmo-Fontanez A, Gautam S, Garcia-Vilanova A, Ye C, Chiem K, Headley C, Dwivedi V, Parodi LM, Alfson KJ, Staples HM, Schami A, Garcia JI, Whigham A, Platt RN 2nd, Gazi M, Martinez J, Chuba C, Earley S, Rodriguez OH, Mdaki SD, Kavelish KN, Escalona R, Hallam CRA, Christie C, Patterson JL, Anderson TJC, Carrion R Jr, Dick EJ Jr, Hall-Ursone S, Schlesinger LS, Alvarez X, Kaushal D, Giavedoni LD, Turner J, Martinez-Sobrido L, Torrelles JB. Lethality of SARS-CoV-2 infection in K18 human angiotensin-converting enzyme 2 transgenic mice. Nat Commun. 2020 Nov 30;11(1):6122. doi: 10.1038/s41467-020-19891-7. PMID 33257679
- [Background] Winkler ES, Bailey AL, Kafai NM, Nair S, McCune BT, Yu J, Fox JM, Chen RE, Earnest JT, Keeler SP, Ritter JH, Kang LI, Dort S, Robichaud A, Head R, Holtzman MJ, Diamond MS. SARS-CoV-2 infection of human ACE2-transgenic mice causes severe lung inflammation and impaired function. Nat Immunol. 2020 Nov;21(11):1327-1335. doi: 10.1038/s41590-020-0778-2. Epub 2020 Aug 24. PMID 32839612
- [Background] Vidal E, Lopez-Figueroa C, Rodon J, Perez M, Brustolin M, Cantero G, Guallar V, Izquierdo-Useros N, Carrillo J, Blanco J, Clotet B, Vergara-Alert J, Segales J. Chronological brain lesions after SARS-CoV-2 infection in hACE2-transgenic mice. Vet Pathol. 2022 Jul;59(4):613-626. doi: 10.1177/03009858211066841. Epub 2021 Dec 27. PMID 34955064
- [Background] Kumari P, Rothan HA, Natekar JP, Stone S, Pathak H, Strate PG, Arora K, Brinton MA, Kumar M. Neuroinvasion and Encephalitis Following Intranasal Inoculation of SARS-CoV-2 in K18-hACE2 Mice. Viruses. 2021 Jan 19;13(1):132. doi: 10.3390/v13010132. PMID 33477869
- [Background] Seehusen F, Clark JJ, Sharma P, Bentley EG, Kirby A, Subramaniam K, Wunderlin-Giuliani S, Hughes GL, Patterson EI, Michael BD, Owen A, Hiscox JA, Stewart JP, Kipar A. Neuroinvasion and Neurotropism by SARS-CoV-2 Variants in the K18-hACE2 Mouse. Viruses. 2022 May 11;14(5):1020. doi: 10.3390/v14051020. PMID 35632761
- [Background] Chen YT, Tsai MS, Yang TL, Ku AT, Huang KH, Huang CY, Chou FJ, Fan HH, Hong JB, Yen ST, Wang WL, Lin CC, Hsu YC, Su KY, Su IC, Jang CW, Behringer RR, Favaro R, Nicolis SK, Chien CL, Lin SW, Yu IS. R26R-GR: a Cre-activable dual fluorescent protein reporter mouse. PLoS One. 2012;7(9):e46171. doi: 10.1371/journal.pone.0046171. Epub 2012 Sep 25. PMID 23049968
- [Background] Leung TF, Wong GW, Hon KL, Fok TF. Severe acute respiratory syndrome (SARS) in children: epidemiology, presentation and management. Paediatr Respir Rev. 2003 Dec;4(4):334-9. doi: 10.1016/s1526-0542(03)00088-5. PMID 14629957
- [Background] Dhochak N, Singhal T, Kabra SK, Lodha R. Pathophysiology of COVID-19: Why Children Fare Better than Adults? Indian J Pediatr. 2020 Jul;87(7):537-546. doi: 10.1007/s12098-020-03322-y. Epub 2020 May 14. PMID 32410003
- [Background] Xie X, Chen J, Wang X, Zhang F, Liu Y. Age- and gender-related difference of ACE2 expression in rat lung. Life Sci. 2006 Apr 4;78(19):2166-71. doi: 10.1016/j.lfs.2005.09.038. Epub 2005 Nov 21. PMID 16303146
- [Background] Consiglio CR, Cotugno N, Sardh F, Pou C, Amodio D, Rodriguez L, Tan Z, Zicari S, Ruggiero A, Pascucci GR, Santilli V, Campbell T, Bryceson Y, Eriksson D, Wang J, Marchesi A, Lakshmikanth T, Campana A, Villani A, Rossi P; CACTUS Study Team; Landegren N, Palma P, Brodin P. The Immunology of Multisystem Inflammatory Syndrome in Children with COVID-19. Cell. 2020 Nov 12;183(4):968-981.e7. doi: 10.1016/j.cell.2020.09.016. Epub 2020 Sep 6. PMID 32966765
- [Background] Miller J, Cantor A, Zachariah P, Ahn D, Martinez M, Margolis KG. Gastrointestinal Symptoms as a Major Presentation Component of a Novel Multisystem Inflammatory Syndrome in Children That Is Related to Coronavirus Disease 2019: A Single Center Experience of 44 Cases. Gastroenterology. 2020 Oct;159(4):1571-1574.e2. doi: 10.1053/j.gastro.2020.05.079. Epub 2020 Jun 4. No abstract available. PMID 32505742
- [Background] Younis JS, Skorecki K, Abassi Z. The Double Edge Sword of Testosterone's Role in the COVID-19 Pandemic. Front Endocrinol (Lausanne). 2021 Mar 16;12:607179. doi: 10.3389/fendo.2021.607179. eCollection 2021. PMID 33796068
- [Background] Mihalopoulos M, Levine AC, Marayati NF, Chubak BM, Archer M, Badani KK, Tewari AK, Mohamed N, Ferrer F, Kyprianou N. The Resilient Child: Sex-Steroid Hormones and COVID-19 Incidence in Pediatric Patients. J Endocr Soc. 2020 Jul 28;4(9):bvaa106. doi: 10.1210/jendso/bvaa106. eCollection 2020 Sep 1. PMID 32864545
- [Background] Mjaess G, Karam A, Aoun F, Albisinni S, Roumeguere T. COVID-19 and the male susceptibility: the role of ACE2, TMPRSS2 and the androgen receptor. Prog Urol. 2020 Sep;30(10):484-487. doi: 10.1016/j.purol.2020.05.007. Epub 2020 May 22. PMID 32620366
- [Background] Cantuti-Castelvetri L, Ojha R, Pedro LD, Djannatian M, Franz J, Kuivanen S, van der Meer F, Kallio K, Kaya T, Anastasina M, Smura T, Levanov L, Szirovicza L, Tobi A, Kallio-Kokko H, Osterlund P, Joensuu M, Meunier FA, Butcher SJ, Winkler MS, Mollenhauer B, Helenius A, Gokce O, Teesalu T, Hepojoki J, Vapalahti O, Stadelmann C, Balistreri G, Simons M. Neuropilin-1 facilitates SARS-CoV-2 cell entry and infectivity. Science. 2020 Nov 13;370(6518):856-860. doi: 10.1126/science.abd2985. Epub 2020 Oct 20. PMID 33082293
- [Background] Mayi BS, Leibowitz JA, Woods AT, Ammon KA, Liu AE, Raja A. The role of Neuropilin-1 in COVID-19. PLoS Pathog. 2021 Jan 4;17(1):e1009153. doi: 10.1371/journal.ppat.1009153. eCollection 2021 Jan. PMID 33395426
- [Background] Bunyavanich S, Do A, Vicencio A. Nasal Gene Expression of Angiotensin-Converting Enzyme 2 in Children and Adults. JAMA. 2020 Jun 16;323(23):2427-2429. doi: 10.1001/jama.2020.8707. PMID 32432657
- [Background] Yang LT, Li WY, Kaartinen V. Tissue-specific expression of Cre recombinase from the Tgfb3 locus. Genesis. 2008 Feb;46(2):112-8. doi: 10.1002/dvg.20372. PMID 18257072